CLINICAL TRIAL: NCT04508946
Title: A Prospective, Randomized Clinical Study Comparing Triple Therapy Regimen to Hydrocortisone Monotherapy in Reducing Mortality in Septic Shock Patients
Brief Title: Triple Therapy in Septic Shock Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Air Force Specialized Hospital, Cairo, Egypt (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019/11
Record Dates: First submitted 2020-08-08; First posted 2020-08-11 (Actual); Last update posted 2021-01-26 (Actual); Status verified 2021-01

CONDITIONS: Septic Shock; Sepsis; Organ Dysfunction Syndrome Sepsis
Keywords: Septic shock; Vitamin C; Thiamine; Hydrocortisone; sepsis
MeSH Terms: conditions — Shock, Septic; Sepsis; Toxemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hydrocortisone Monotherapy (Active Comparator): Hydrocortisone Monotherapy
  Interventions: Drug: vitamin c - thiamine- hydrocortisone
- triple therapy regimen (vitamin c - thiamine- hydrocortisone) (Experimental): triple therapy regimen (vitamin c - thiamine- hydrocortisone)
  Interventions: Drug: vitamin c - thiamine- hydrocortisone

INTERVENTIONS:
Drug: vitamin c - thiamine- hydrocortisone — Triple therapy regimen (vitamin c - thiamine- hydrocortisone)
  Other Names: Triple therapy

SUMMARY:
this study is conducted to evaluate the role of the novel triple therapy combination in reducing the mortality rate, reducing the shock time, and reversal of organ damage.

the study includes two arms, the first arm is the control which received hydrocortisone monotherapy and the second arm is the intervention arm which received the triple therapy regimen.

calculation of 28 days in-hospital mortality is the primary outcome. shock time, vasopressor doses, infection markers, and organ function tests are the secondary outcomes.

the data will be analyzed by student t-test or Mann Whitney test, Fischer exact or chi-square test for numbers, repeated measures ANOVA will be used to consider confounders and other parameters, mortality will be expressed by Kaplan Meier and ROC curve.

For Multivariate analysis of repeated quantitative outcomes, linear mixed models were used to quantify the relationship between one dependent variable (SOFA, SCr, doses of vasopressors) and many independent variables including group type and sepsis phenotype adjusted to other clinical and demographic factors.

DETAILED DESCRIPTION:
Background:

"Sepsis" is a life-threatening organ dysfunction caused by the dysregulated host response to infection. Septic Shock: Subset of sepsis with circulatory and cellular/metabolic dysfunction associated with a higher risk of mortality. Organ dysfunction can be identified by acute change in the total Sequential Organ Failure Assessment (SOFA) score of 2 points or higher consequent to the infection.

Septic shock patients can be identified by developing sepsis with persistent arterial hypotension requiring vasopressors to keep mean arterial pressure (MAP) above 65 mm Hg and having serum lactate above 2 mmol/L. In hospitals, the mortality of septic shock according to retrospective studies is around 35%-54%. Pneumonia is the most common site of infection (about 50%) of cases, followed by intra-abdominal infection and urinary tract infection.

The (1-hr Bundle) is the cornerstone of the management, it encourages clinicians to act as quickly as possible to obtain blood cultures, administer broad-spectrum antibiotics, start appropriate fluid resuscitation, measure lactate, and begin vasopressors if clinically indicated. Ideally, these interventions would all begin in the first hour from sepsis recognition but may not necessarily be completed in the first hour. However, over the last few years, there have been interesting investigational novel therapeutic approaches. One of them is the use of high dose vitamin C. A small retrospective study demonstrated a mortality benefit by using high dose vitamin C, thiamine (vitamin B1), and hydrocortisone (Triple therapy) for treatment of septic shock in the adult population.

The normal plasma vitamin C level is ≥ 23 µmol/l. A recent study found that 88% of septic shock patients have hypovitaminosis C (<23 µmol/l), while 38% have a scurvy level (<11 µmol/l). The acute deficiency of vitamin C in this category of patients may be caused by the increased metabolic consumption due to critical illness such (trauma, burn, septic shock, etc.).

Vitamin C has pleiotropic effects such as antioxidant (direct radical scavenger- reduction of reactive oxygen species (ROS) production-regeneration of antioxidants), anti-inflammatory, and immune-supporting, cofactor/co-substrate biosynthesis, increasing catecholamine sensitivity and protection of microcirculation. Vitamin C enteral intake is insufficient in critically ill patients due to saturable mucosal sodium-dependent vitamin C transporter 1 (SCVC1). So, supplementation of high doses of vitamin C by intravenous route can restore normal plasma concentration and reverse the stress and its sequences (reduce the incidence of organ failure, reduce vasopressor support, and may reduce the overall mortality).

Recent small controlled studies suggested the dosing range of vitamin C is from 6-16 gm/day. Also, a dose-response relationship in patients who received high doses of vitamin C was proven. Vitamin C is actively transported in tissue cells by (SCVC2), leading to achieving a high intracellular level than the plasma especially in leukocytes and neurons protecting them against ROS. While high doses of vitamin C given were not associated with any harms related to the drug, there is a theoretical concern regarding the use of high doses related to the potential risk for developing oxalate crystals in the urinary tract, For this reason, co-administration of thiamine with these high doses of vitamin C acts as a co-enzyme for the function of glyoxalate-amino transferase which catalyzes the degradation of glyoxalate to carbon dioxide instead of the oxalate. Another note is a short course of high doses vitamin C has not been found to increase the risk of renal calculi in the previous studies. Also, patients with glucose-6-phosphate dehydrogenase (G6PD) enzyme deficiency are at risk of hemolysis with high doses of vitamin C.

Thiamine has a crucial role in cellular metabolic processes. Thiamine deficiency is common in critically ill patients when becomes insufficient pyruvate not converted to acetyl coenzyme A resulting in impaired aerobic respiration and switch to anaerobic respiration leading to elevate of lactate level. Previous studies showed improvement in lactate level and in organ dysfunction with supplementation of thiamine for critically ill patients, thiamine dose is 200mg every 12 hours.

Hydrocortisone is another major component of the recommended triple therapy, the dose of hydrocortisone in septic shock is 200 mg/day, The rationale for its use is that, in septic shock, the released component of the cell membrane of gram-negative and gram-positive bacteria and endotoxins induce nitric oxide synthase which promotes the relaxation of vascular beds in addition to releasing of inflammatory cytokines such tumor necrosis factor (TNF-alpha) and interleukins (IL-1). These cytokines suppress the action of Adreno-Cortico Trophic Hormone (ACTH) on the adrenal gland and decrease the endogenous cortisol and compete with cortisol on receptor sites and diminish its effect, By supplying hydrocortisone, reversing of these mechanisms occurs which improves response to vasopressors, blocks phospholipase A2 then reduces prostacyclins and prostaglandins (vasodilators), reducing the diminished steroid action at receptor sites. Synergism appears between hydrocortisone and vitamin C based on two roles, one of them is glucocorticoid binding to glucocorticoid receptors is negatively affected by oxidizing molecules and this can be reversed by administration of high doses of vitamin C which restores the glucocorticoid receptor functions.

Also, it was found that the transcellular transportation of vitamin C via SVCT2 is impaired due to the downregulation of this transporter during septic shock, hydrocortisone has been shown increasing the expression of this transporter and then increases the cellular uptake.

Aim of the study To determine the effectiveness of triple therapy regimen (vitamin C, vitamin B1, and Hydrocortisone) in the reduction of mortality of septic shock patients.

Methodology Study subjects and designs This is an interventional, controlled, single-blind prospective parallel study to be conducted in the (ICUs) at the Air Force Specialized Hospital (AFSH), Cairo, Egypt.

Subjects will be selected according to the following inclusion and exclusion criteria:

Sample size Sample size will be calculated based on this equation

assuming the following parameters: Anticipated Incidence of mortality: GP1 (hydrocortisone arm) = 40.4%, in GP 2 (triple therapy arm) = 8.5%.

Alpha = 0.05, power = 95%, enrollment ratio = 1 So each group will consist of 44 patients (total = 88).

* By considering dropout rate = 20%, So each group will consist of 53 patients and the total sample size =106 patients.
* The first arm will take the triple therapy regimen (vitamin C, vitamin B1, and Hydrocortisone), the Second arm will take Hydrocortisone as the standard of care.

Data collection:

From each patient the following data will be collected:

* Age, gender, height and weight, and any allergies (on admission)
* Causes of ICU admission (on admission).
* Patient's past medical history (PMH) (on admission)
* SOFA score to be assessed on admission and daily (primary outcome) [28] and Acute Physiologic Assessment and Chronic Health Evaluation (APACHE ӏӏ) [29] score (on admission only).
* Hemodynamic data (blood pressure, pulse, central venous pressure (CVP), respiratory rate, O2 saturation) on admission, and daily.
* Infection markers (total leukocytic count, CRP), lactate level, serum creatinine, Aspartate Aminotransferase (AST), Alanine aminotransferase (ALT). on admission and for follow- up daily (secondary outcome).

Statistical analysis

Different statistical tests selection will be based on the type of data and the calculated outcome:

* Mortality (primary outcome) calculation will be evaluated by the chi-square test.
* Reversal of organs failure, weaning from the mechanical ventilator, and vasopressors will be evaluated using the Mann-Whitney test.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years.
* Diagnosis of septic shock has been established (need vasopressors to maintain MAP ≥ 65, lactate ≥ 2mmol/L and SOFA score ≥2) [25,26].

Exclusion Criteria:

* Pregnancy and lactation.
* Refusal of attending staff or patient family.
* Contraindication to any of the components of the triple therapy regimen such as (hypersensitivity to vitamin C and Patients with G6PD deficiency).
* Patients on immunosuppressive medications and oncology patients. Do not resuscitate/do not intubate (DNR, DNI) patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2020-11-09 (Actual); Study Completion 2020-11-09 (Actual)

PRIMARY OUTCOMES:
The number of patients who died within 28 days. | 28 days
  patients were followed up daily for 28 days, this is the number of patients who died within 28 days.
ICU Mortality | Within 28 days
  The number of patients who died during ICU stay

SECONDARY OUTCOMES:
the number of days that are needed to off the patients from vasopressors. | 28 Days
  average number of days that are needed to off the patients from vasopressors.
the number of days that are needed to off the patients from mechanical ventilation. | 28 days
  average number of days that are needed to off the patients from mechanical ventilation.
Change in organ's functions test such as (serum creatinine, Alanine Aminotransferase (ALT) | 28 days
  change was calculated as the values at ICU stay and specific cut off points (after 48 hr, after 96 hr).

CONTACTS AND LOCATIONS:
Overall Officials: Abdelrhman Hussein, Principal Investigator — Air Force Specialized Hospital
Locations (1):
- Air Force Specialized Hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Dellinger RP, Levy MM, Rhodes A, Annane D, Gerlach H, Opal SM, Sevransky JE, Sprung CL, Douglas IS, Jaeschke R, Osborn TM, Nunnally ME, Townsend SR, Reinhart K, Kleinpell RM, Angus DC, Deutschman CS, Machado FR, Rubenfeld GD, Webb SA, Beale RJ, Vincent JL, Moreno R; Surviving Sepsis Campaign Guidelines Committee including the Pediatric Subgroup. Surviving sepsis campaign: international guidelines for management of severe sepsis and septic shock: 2012. Crit Care Med. 2013 Feb;41(2):580-637. doi: 10.1097/CCM.0b013e31827e83af. PMID 23353941
- [Result] Plevin R, Callcut R. Update in sepsis guidelines: what is really new? Trauma Surg Acute Care Open. 2017 Sep 7;2(1):e000088. doi: 10.1136/tsaco-2017-000088. eCollection 2017. PMID 29766091
- [Result] Korosec Jagodic H, Jagodic K, Podbregar M. Long-term outcome and quality of life of patients treated in surgical intensive care: a comparison between sepsis and trauma. Crit Care. 2006;10(5):R134. doi: 10.1186/cc5047. PMID 16978417
- [Result] Zahar JR, Timsit JF, Garrouste-Orgeas M, Francais A, Vesin A, Descorps-Declere A, Dubois Y, Souweine B, Haouache H, Goldgran-Toledano D, Allaouchiche B, Azoulay E, Adrie C. Outcomes in severe sepsis and patients with septic shock: pathogen species and infection sites are not associated with mortality. Crit Care Med. 2011 Aug;39(8):1886-95. doi: 10.1097/CCM.0b013e31821b827c. PMID 21516036
- [Result] Angus DC, van der Poll T. Severe sepsis and septic shock. N Engl J Med. 2013 Aug 29;369(9):840-51. doi: 10.1056/NEJMra1208623. No abstract available. PMID 23984731